CLINICAL TRIAL: NCT01310127
Title: Clinical Outcomes of Bromday (Bromfenac Ophthalmic Solution) 0.09% QD vs. Nevanac (Nepafenac Ophthalmic Suspension) 0.1% TID for Treatment of Ocular Inflammation Associated With Cataract Surgery
Brief Title: Clinical Outcomes of Bromday (Bromfenac Ophthalmic Solution) 0.09% QD vs. Nevanac (Nepafenac Ophthalmic Suspension) 0.1%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Toyos Clinic (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Melissa Toyos, Principal Inevstigator, Toyos Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAC-02-11
Record Dates: First submitted 2011-03-01; First posted 2011-03-08 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Inflammation; Pseudophakia
Keywords: NSAID; Ocular Inflammation; bromfenac
MeSH Terms: conditions — Inflammation; Pseudophakia | interventions — bromfenac; nepafenac

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bromday (Experimental): Patients receiving Bromday self-administered one drop of bromfenac 0.09% daily as a topical ophthalmic drop three days prior to cataract surgery, on the day of cataract surgery and 21 days post operatively.
  Interventions: Drug: Bromfenac
- Nevanac (Active Comparator): Patients in this arm self-administered nepafenac topical ophthalmic drops three times daily beginning 3 days prior to cataract surgery, on the day of surgery and for 21 days postoperatively in addition to usual cataract procedure.
  Interventions: Drug: Nepafenac

INTERVENTIONS:
Drug: Bromfenac — bromfenac 0.9% QD starting 3 days prior to cataract surgery, on the day of surgery and for up to 45 days after surgery
  Other Names: Bromday (bromfenac ophthalmic solution) 0.9%
  Arms: Bromday
Drug: Nepafenac — nepafenac ophthalmic suspension 0.1% TID dosed 3 days prior to cataract surgery, on the day of surgery, and for up to 45 days after surgery
  Other Names: Nevanac (nepafenac ophthamic suspension) 0.1%
  Arms: Nevanac

SUMMARY:
This is a single-center, randomized, investigator-masked, parallel group, and active-comparator controlled study investigating the clinical outcomes for visual acuity and macular thickness after treatment with Bromday (bromfenac ophthalmic solution) 0.09% QD or Nevanac (nepafenac ophthalmic suspension) 0.1% TID in subjects who have undergone cataract extraction with posterior chamber intraocular lens implantation.

DETAILED DESCRIPTION:
Two topical NSAIDs currently approved for postoperative treatment of pain and inflammation in cataract surgery are bromfenac 0.09% and nepafenac 0.1%. Both purport to treat ocular inflammation by acting as a potent inhibitor of COX-1 and COX-2 enzymes. Clinical studies to date lack clarity on which topical NSAID may be the most efficacious.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female at least 18 years of age who are scheduled for unilateral cataract surgery (phacoemulsification or extracapsular) with posterior chamber intraocular lens implantation and for whom no other ophthalmic surgical procedures (e.g., relaxing incisions, iridectomy, conjunctival excisions, etc) are to be conducted during the cataract surgery.
* Agree not to have any other ocular surgical procedures in the study or fellow (non study) eye within 15 days prior to the initiation of dosing with the test article or throughout the duration of the study.
* Have a Best Corrected Visual Acuity of 20/200 or better in either eye.
* If a woman capable of becoming pregnant, agree to have urine pregnancy testing performed at screening (must be negative) and agree to use a medically acceptable form of birth control throughout the study duration and for at least one week prior to and after completion of the study. Women considered capable of becoming pregnant include all females who have experienced menarche and who have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy).
* Have IOP ≥ 5 mmHg and ≤ 22 mmHg (in study eye) with or without anti glaucoma therapy at the pre operative screening visit (if >22 mmHg, adjust following pachymetry).

Exclusion Criteria:

* Have known hypersensitivity to bromfenac or Nepafenac or to any component of the test article (including "procedural" medications such as anesthetic and/or fluorescein drops, dilating drops, etc.).
* Have a known hypersensitivity to salicylates (i.e., aspirin) or to other non steroidal anti inflammatory drugs (NSAIDs).
* Have intraocular inflammation (i.e., cells or flare in the anterior chamber as measured on slit lamp examination) in the study eye at the screening visit.
* Have a known blood dyscrasia or bone marrow suppression, a diagnosis of uncontrolled/unstable peptic ulcer disease, inflammatory bowel disease, or ulcerative colitis, or any uncontrolled/unstable pulmonary, cardiac, vascular, autoimmune, hepatic, renal, or central nervous system disease.
* Have used ocular, topical, or systemic NSAIDs or ocular, topical, or systemic gentamicin, or cyclosporine ophthalmic emulsion within 7 days prior to initiation of dosing with the test article or throughout the duration of the study.
* Have used any ocular prostaglandins within 30 days prior to initiation of dosing with the test article or throughout the duration of the study.
* Have active corneal pathology noted in the study eye at the screening visit. Active corneal pathology is defined as corneal pathology that is non stable, or greater than mild, or will compromise assessment of the safety or efficacy of treatment. Superficial punctate keratitis in the study eye is a criterion for exclusion.
* Have used topical, ocular, inhaled or systemic steroids within 14 days prior to screening.
* Have had radial keratotomy, corneal transplant, or corneal refractive surgery in the study eye within the last two years.
* Are pregnant or nursing/lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Cable, MD, Principal Investigator — Discover Vision Centers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical outcomes of bromfenac ophthalmic solution 0.09% QD and nepafenac 0.1% ophthalmic suspension TID post cataract surgery with posterior chamber intraocular lens implantation, specifically looking at any differences in Early Treatment Diabetic Retinopathy Study visual acuities, macular volume, and/or retinal thickness changes.
Pre-assignment Details: Subjects were randomized to receive bromfenac(n=12) QD or nepafenac(n=11) TID. Dosing was 3 days before cataract surgery through day 21 postop. Subjects could not have used ocular/topical, systemic NSAIDs, gentamicin, or cyclosporine ophthalmic emulsion 7 days or prostaglandins 30 days prior to initial dosing of test article or during the study.
Groups:
- Bromday: Bromfenac : bromfenac 0.9% QD starting 3 days prior to cataract surgery, on the day of surgery and for up to 45 days after surgery
- Nevanac: Nepafenac : nepafenac ophthalmic suspension 0.1% TID dosed 3 days prior to cataract surgery, on the day of surgery, and for up to 45 days after surgery
Period: Overall Study
Arm/Group | Bromday | Nevanac
Started | 12 | 11
Completed | 10 | 10
Not Completed | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — advanced psc cataract outlier | 1 | 0

BASELINE CHARACTERISTICS:
Population: 1 nepafenac patient did not use test article prior to surgery. 1 bromday patient used nsaid during study. 1 bromday patient had advanced psc cataract.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bromday | Nevanac | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (10.5) | 69.7 (9.0) | 69.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuities
Description: ETDRs visual acuities measured at week 6 following uncomplicated phacoemulsification (phaco). ETDRS charts are a standardized eye chart for visual acuity testing accepted by the National Eye Institute and the Food and Drug Administration. The scale is 30-90 letters with higher numbers signifying improved visual acuities.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Bromday | Nevanac
Number analyzed (Participants) | 10 | 10
letters | 51.3 (6.818) | 52 (6.750)

2. Primary Outcome: Summed Ocular Inflammation Score (SOIS)
Description: An assessment of the cells and flare, signs of inflammation in ocular tissue. SOIS (summed ocular inflammation) = cells in the anterior chamber/1mmx1mm high powered field+flare/1mmx1mm high powered field. The score of the number of cells in the anterior chamber per 1mmx1mm high powered field ranges from 0-4: 0=no cells, 1=1-5 cell, 2=6-15 cells, 3=16-30 cells, 4>=30 cells.Flare scores range from 0-3:(0=none, 1=mild, 2=moderate, 3=severe). Cell+flare are added together (cell score + flare score=SOIS score) for a SOIS score (minimum score=0 and maximal score of 7). Higher numbers would indicate more inflammation.The SOIS scale could range from 0-7 with 0 indicating no cells, no flare and 7 reflecting maximal cell 4(>30 cell/high powered field +3 (severe flare).
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bromday | Nevanac
Number analyzed (Participants) | 10 | 10
units on a scale | 0.15 (0.229) | 0.2 (0.245)

3. Primary Outcome: OCT Retinal Thickness
Description: Stratus OCT scan retinal thickness/volume tabular output report. An experienced ophthalmic technician obtained two scan patterns. The first was the fast macular thickness using 6 radial line scans through a common central axis (fovea) with a retinal thickness/volume tabular output and a retinal-thickness output report. Central retinal thickness was defined as the distance between the inner limiting membrane of the retina and the inner border of the choriocapillaris in the central 1 mm area of the minimum 7 mm posterior pole scan. All scans were reviewed by the principal investigator for quality of foveal centration and signal strength. Macular volume is an objective indicator of macualr swelling and can illustrate the amount of inflammation following surgery. Only the study eye was assessed.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: micrometers cubed
Arm/Group | Bromday | Nevanac
Number analyzed (Participants) | 10 | 10
micrometers cubed | 230.7 (30.63) | 223.8 (25.36)

4. Primary Outcome: Macular Volume
Description: Stratus OCT by experienced technician. Reviewed by principal investigator for quality of foveal centration and signal strength
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: mm cubed
Arm/Group | Bromday | Nevanac
Number analyzed (Participants) | 10 | 10
mm cubed | 0.1815 (0.49) | 0.1765 (0.34)

ADVERSE EVENTS:
Arm/Group | Bromday | Nevanac
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bromday (N=12) | Nevanac (N=11)
recurrent symptomatic postoperative iritis (Eye disorders) | 0 (0) | 1 (1) — symptomatic recurrent postoperative iritis at final postoperative visit necessitating topical rescue medications

LIMITATIONS AND CAVEATS:
The major limitation in the study is that it was a small pilot study so that the direct correlations of the study variable could not be evaluated. There were ethnic differences in the groups that could also influence the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No